CLINICAL TRIAL: NCT04640103
Title: An Observational Study Evaluating the Safety and Effectiveness of Perioperative Immunotherapy in Microsatellite Instability-high Gastrointestinal Tumors
Brief Title: An Observational Study of Perioperative Immunotherapy in MSI-H Gastrointestinal Tumors
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shen Lin (Other)
Responsible Party: Sponsor-Investigator, Shen Lin, Professor, Peking University
Organization: Peking University (Other)
Other Study IDs: MSI Perioperative ICI
Record Dates: First submitted 2020-11-16; First posted 2020-11-23 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: To Evaluate the Safety and Effectiveness of Immunotherapy During the Perioperative Treatment Stage in MSI-H Gastrointestinal Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- adjuvant therapy: Patients who received immunotherapy in adjuvant treatment stage only
  Interventions: Other: No interventions
- neoadjuvant therapy: Patients who received immunotherapy in neoadjuvant treatment stage and achieved R0 resection
  Interventions: Other: No interventions

INTERVENTIONS:
Other: No interventions — No interventions

SUMMARY:
Gastrointestinal cancer like Gastric cancer and colorectal cancer are high-incidence tumors worldwide. Surgery is the only curable way. Perioperative treatment can improve the survival of patients. Microsatellite instability-high（MSI-H）are a special subtype of gastrointestinal tumors, accounting for about 15-22%. According to current research, patients with this type of gastrointestinal tumors cannot benefit from traditional perioperative chemotherapy, which directly affects the long-term survival of patients. Because patients with MSI-H have a unique tumor immune microenvironment, thus they are more likely to benefit from immunotherapy. Current studies have confirmed that the use of immunotherapy during palliative care can prolong the survival of patients with MSI-H. In the neoadjuvant treatment stage, according to the previous clinical practice of our center, the use of immunotherapy can make some patients achieve complete postoperative pathological remission. However, in the perioperative treatment stage, the value of immunotherapy is still lack of powerful clinical evidence.

Based on this, our group intends to start an observational study to prospectively enroll patients with MSI-H gastrointestinal tumor using immunotherapy during the perioperative period.The primary endpoint is safety while survival outcomes as secondary endpoints. In order to evaluate the safety and effectiveness of immunotherapy during the perioperative treatment stage in MSI-H gastrointestinal cancer

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old,diagnosed as gastric or colorectal cancer by pathology;
2. Diagnosed as a mismatch repair deficient by immunohistochemistry,or diagnosed as microsatellite instability-high by polymerase chain reaction(PCR) or next-generation sequencing(NGS);
3. Suitable for tumor radical resection;
4. Join this trial voluntarily,and could sign an informed consent form;
5. With good compliance.

Exclusion Criteria:

1. Do not use immunotherapy containing PD-1/PD-L1 antibody during the perioperative period;
2. Simultaneous diagnosis of dual primary tumors, and the second tumor cannot be resected radically, or the second tumor is not dMMR/MSI-H;
3. Complicate with uncontrollable immune system diseases;
4. Patients who need to use glucocorticoids and other immunosuppressive agents for a long time;
5. Patients who received live vaccines or live attenuated vaccines within 30 days before the medication, except for inactivated vaccines;
6. Those who cannot provide detailed medical records or cannot cooperate with follow-up.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Outpatients and inpatients in Beijing Cancer Hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse event rate | Up to 1 years
  Safety

SECONDARY OUTCOMES:
Overall survival | Up to 5 years
  From the time of enrollment to death caused by any reason
Disease-free survival | Up to 3 years
  From the time of enrollment to disease recurrence or death caused by any reason
Incidence of second tumor in patients with Lynch syndrome | Up to 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China